CLINICAL TRIAL: NCT04533165
Title: Feasibility and Effectiveness of an Innovative Exercise Program to Reduce Fatigue in Rural Cancer Survivors
Brief Title: Virtual Exercise Program to Reduce Cancer Related Fatigue
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cancer League of Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-2015.cc
Record Dates: First submitted 2020-08-06; First posted 2020-08-31 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Cancer; Cancer-related Problem/Condition; Fatigue
Keywords: Exercise; Telehealth; Cancer-related fatigue
MeSH Terms: conditions — Neoplasms; Fatigue; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm pilot interventional trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual exercise program (Experimental): This arm will receive the virtual exercise program.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 12 week exercise prescription targeting 3 days of at least 30 min of aerobic exercise and 2 days of resistance exercise per week. Adapted to individual abilities, goals, and needs. Exercise intensity targets a 6-7 out of 10 on a 0-10 rate of perceived exertion scale.

SUMMARY:
The objective of this investigation is to establish the feasibility and initial effectiveness of a novel exercise program for rural cancer survivors in Colorado suffering from cancer related fatigue. Participation in an exercise program has regularly been shown to reduce fatigue in cancer survivors, though in-person, supervised participation has a greater effect on fatigue than home-based programs with no supervision. Access to these supervised programs are limited in rural areas, restricting the ability of rural cancer survivors to experience the fatigue-reducing benefits of exercise. The proposed program will use information on improvements in fatigue from participants in the BfitBwell Cancer Exercise Program to monitor improvements in fatigue in rural cancer survivors performing a home exercise program and trigger a telehealth session with a cancer exercise specialist to adapt the exercise prescription when improvements are less than expected. The BfitBwell Program is an established exercise program at the Anschutz Health and Wellness Center which has worked with over 600 cancer survivors and is highly effective at reducing cancer related fatigue. The goal of the program is to replicate the effects of a successful supervised exercise program in rural cancer survivors who do not have access to this type of program. This investigation will recruit 20 rural cancer survivors experiencing fatigue and assess their ability to participate in the program, as well as how well the program improves their fatigue. Interviews will be conducted with participants after the program to determine how future versions of the program could be improved. The investigators anticipate that this program will be feasible and effective, providing preliminary data to pursue a large-scale clinical trial of the program following this project's completion.

DETAILED DESCRIPTION:
The proposed exercise program utilizes a novel reference chart system to monitor cancer-related fatigue (CRF) and trigger necessary interventions. This reference chart has been developed from CRF data collected in 173 cancer survivors participating in the BfitBwell Program, a highly effective supervised exercise program pioneered at the University of Colorado. The reference chart estimates the continuous trajectory of fatigue improvement during the three-month program. The focus of this study is to extend the benefits of an effective, supervised exercise program to rural Coloradoans via a home exercise program supported by CRF monitoring and symptom-triggered telehealth sessions. Deviations from estimated improvements in CRF will trigger telehealth sessions with a cancer exercise specialist (CES) to adapt the exercise prescription, in real time, as in a supervised program. The intent is to replicate the effects of a supervised exercise program in cancer survivors in rural areas without access to such programs. The feasibility, effectiveness, and design of the program will be assessed with two specific aims.

Aim 1: Determine the feasibility and preliminary effectiveness of the proposed exercise program.

Objective 1a: Assess the enrollment rate of patients able and willing to participate in the program and the adherence of patients enrolled in the program to their prescribed exercise, CRF monitoring, and telehealth session participation.

Objective 1b: Assess the effect of the proposed program on CRF improvements in enrolled participants and compare this effect to that of the supervised BfitBwell exercise program.

Exploratory Objective 1: Assess the feasibility of the semi-continuous remote monitoring of fatigue (ecological momentary assessment) to better tailor the program to more acute changes in CRF.

Aim 2: Assess participant perspectives of barriers and facilitators to participation in the prescribed exercise and CRF monitoring.

Objective 2: Gather qualitative data on barriers and facilitators to participation from all participants enrolling in the program using semi-structured interviews.

This is an innovative program, being the first exercise intervention to implement real time adaptations for rural patients, with decisions anchored against a novel symptom monitoring system. Qualitative data will be collected to improve the next iteration of the program and to inform a future, large-scale clinical trial of program implementation in rural populations. The long-term goal is to develop a feasible and effective exercise program for rural cancer survivors which replicates the benefits of supervised exercise programs to which access may be restricted in rural settings.

This is a prospective, single-arm pilot intervention trial. It will collect objective data on the feasibility and effectiveness of the intervention, as well as qualitative data to inform how the intervention could be improved in future iterations. The exploratory aim will collect data on "in-the-moment" fatigue that could also inform novel future versions of the intervention.

This investigation will recruit adult cancer survivors treated at the University of Colorado Cancer Center (aged 18 years and over) who live in rural Colorado, have completed cancer treatment, and report moderate-to-severe CRF (> 3 on a 0-10 scale, per NCCN definition). Cancer type will be limited to the three types with the highest anticipated new cases in Colorado in 2020: breast, prostate, and lung. Only survivors who have completed medical treatment (chemotherapy and/or radiation), with curative intent, within the past 12 months, and have no additional treatment planned for the next four months, will be recruited. Rural participants will be defined as those who have greater than a 1-hour commute to the major front range cities (Denver, Fort Collins, and Colorado Springs). Participants must have home internet access and smartphones to allow participation in telehealth sessions and remote monitoring of exercise participation and fatigue. Participants with medical conditions that would impact the safety of, or participation in, an exercise program will be excluded. Twenty participants will be recruited in one year, with the goal of retaining at least 15 through the final assessment.

Participants will complete assessments (baseline and final) and exercise sessions virtually. The primary outcome measure will be the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) scale. Other assessment items will include measures of physical fitness and function. CRF will be assessed by questionnaires every two weeks, and semi-continuously with a smartphone application. The exercise program is 12 weeks long, and includes 2 mandatory virtual exercise sessions, and up to 5 triggered virtual exercise sessions. Participants will be mailed equipment to complete the study upon enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>= 18 years) cancer survivor.

  * A maximum age of 80 will be set as virtual exercise may become unsafe as individuals get older.
* A cancer diagnosis of any type

  * CRF is a common symptom across cancer types and the current CRF reference chart was developed using data from patients with all cancer types.
* Current report of moderate-to-severe fatigue (> 3 on a 0-10 scale, per NCCN definition31)
* Live in rural Colorado and surrounding areas (> 1-hour commute to major front range city [Denver, Fort Collins, and Colorado Springs])

  * This program attempts to target individuals in Colorado and surrounding areas with restricted access to fitness centers that may offer cancer specific services, most likely found in major front range cities. We have defined rural in terms of commute time to these cities, as it is the commute to these centers that restricts access.
* Completed medical cancer treatment (chemotherapy and/or radiation) with curative intent within past 12 months or currently on treatment with no planned changes for the next 4 months (e.g. maintenance or palliative therapy).

  * No additional treatment planned for next 4 months.
  * These restrictions are made to ensure the validity of tracking changes with the established reference chart, which was developed using data from cancer survivors who had recently completed therapy or were on therapy14. It is unclear how fatigue response to exercise may change in survivors further out from treatment completion.
* High-speed home internet and smartphone (or laptop with camera).

Exclusion Criteria:

- Medical conditions that would impact the safety of, or participation in, an exercise program. This includes:

* Orthopedic conditions such as advanced osteoarthritis, mobility-limiting amputations or chronic injuries, or mobility- limiting acute orthopedic injuries
* Advanced rheumatoid arthritis
* Widespread chronic pain conditions such as fibromyalgia
* Significant balance impairment increasing the risk of falling
* Pulmonary conditions such as chronic obstructive pulmonary disease, emphysema, interstitial lung disease, use of supplemental oxygen
* Known cardiovascular disease, uncontrolled hypertension, or new cardiac event within the past 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) at 12 weeks | Baseline (week 0), 12 weeks
  13-item instrument widely used to assess cancer related fatigue. Score range: 0-52. Lower scores indicate more fatigue.

SECONDARY OUTCOMES:
Changes in Steps per day | Baseline (week 0), 12 weeks
  Average steps per day over a 7 day period, assessed with commercial fitness tracker
Changes in Average sleep time | Baseline (week 0), 12 weeks
  Average sleep time per day over a 7 day period, assessed with commercial fitness tracker
Changes in Single limb stance | Baseline (week 0), 12 weeks
  Time participant can stand on one leg, up to 30 s
Changes in Gait speed | Baseline (week 0), 12 weeks
  Gait speed over a 4 m distance, in m/s
Changes in Timed up and go | Baseline (week 0), 12 weeks
  Time (in s) to rise from a chair, walk 3 m, turn around, walk back to chair, and sit down
Changes in 30 s Sit-to-Stand | Baseline (week 0), 12 weeks
  Number of times one can stand and sit from a chair in 30 s
Changes Tecumseh Step Test | Baseline (week 0), 12 weeks
  Participants steps on and off an 8" step at a rate of 24 steps/min for 3 min. Heart rate is recorded at 30 s and 1 min after completion.
Changes in Functional Assessment of Cancer Therapy-General form (FACT-G) at 12 weeks | Baseline (week 0), 12 weeks
  Common questionnaire assessing health related quality of life in cancer survivors, range 0-108, higher scores indicate better quality of life
Changes in Functional Assessment of Cancer Therapy-General form (FACT-G) at 6 month | Baseline (week 0), 6 months
  Common questionnaire assessing health related quality of life in cancer survivors, range 0-108, higher scores indicate better quality of life
Changes in Functional Assessment of Cancer Therapy-General form (FACT-G) at 9 months | Baseline (week 0), 9 months
  Common questionnaire assessing health related quality of life in cancer survivors, range 0-108, higher scores indicate better quality of life
Changes in Functional Assessment of Cancer Therapy-General form (FACT-G) at 15 months | Baseline (week 0), 15 months
  Common questionnaire assessing health related quality of life in cancer survivors, range 0-108, higher scores indicate better quality of life
Changes in Multidimensional Fatigue Inventory (MFI) at 12 weeks | Baseline (week 0), 12 weeks
  Questionnaire with multiple subscales of fatigue identified. Score range: 0-100, higher scores indicate increased fatigue
Changes in Multidimensional Fatigue Inventory (MFI) at 6 months | Baseline (week 0), 6 months
  Questionnaire with multiple subscales of fatigue identified. Score range: 0-100, higher scores indicate increased fatigue
Changes in Multidimensional Fatigue Inventory (MFI) at 9 months | Baseline (week 0), 9 months
  Questionnaire with multiple subscales of fatigue identified. Score range: 0-100, higher scores indicate increased fatigue
Changes in Multidimensional Fatigue Inventory (MFI) at 15 months | Baseline (week 0), 15 months
  Questionnaire with multiple subscales of fatigue identified. Score range: 0-100, higher scores indicate increased fatigue
Changes in Hospital Anxiety and Depression Scale (HADS) at 12 weeks | Baseline (week 0), 12 weeks
  Questionnaire to assess anxiety and depression in populations with medical conditions. Score range: 0-42, higher scores indicate presence of anxiety and depression
Changes in Hospital Anxiety and Depression Scale (HADS) at 6 months | Baseline (week 0), 6 months
  Questionnaire to assess anxiety and depression in populations with medical conditions. Score range: 0-42, higher scores indicate presence of anxiety and depression
Changes in Hospital Anxiety and Depression Scale (HADS) at 9 months | Baseline (week 0), 9 months
  Questionnaire to assess anxiety and depression in populations with medical conditions. Score range: 0-42, higher scores indicate presence of anxiety and depression
Changes in Hospital Anxiety and Depression Scale (HADS) at 15 months | Baseline (week 0), 15 months
  Questionnaire to assess anxiety and depression in populations with medical conditions. Score range: 0-42, higher scores indicate presence of anxiety and depression
Change in Godin Leisure-Time Physical Activity Questionnaire (GLTPAQ) at 12 weeks | Baseline (week 0), 12 weeks
  Self-report of time spent in light, moderate, and vigorous physical activity in minutes.
Change in Godin Leisure-Time Physical Activity Questionnaire (GLTPAQ) at 6 months | Baseline (week 0), 6 months
  Self-report of time spent in light, moderate, and vigorous physical activity in minutes.
Change in Godin Leisure-Time Physical Activity Questionnaire (GLTPAQ) at 9 months | Baseline (week 0), 9 months
  Self-report of time spent in light, moderate, and vigorous physical activity in minutes.
Change in Godin Leisure-Time Physical Activity Questionnaire (GLTPAQ) at 15 months | Baseline (week 0), 15 months
  Self-report of time spent in light, moderate, and vigorous physical activity in minutes.
Change in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) at 6 months | Baseline (week 0), 6 months
  13-item instrument widely used to assess cancer related fatigue. Score range: 0-52. Lower scores indicate more fatigue.
Change in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) at 9 months | Baseline (week 0), 9 months
  13-item instrument widely used to assess cancer related fatigue. Score range: 0-52. Lower scores indicate more fatigue.
Change in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) at 15 months | Baseline (week 0), 15 months
  13-item instrument widely used to assess cancer related fatigue. Score range: 0-52. Lower scores indicate more fatigue.

OTHER OUTCOMES:
Ecological momentary assessments of fatigue | Semi-continuous throughout program, up to 12 weeks
  11 point fatigue intensity scale with higher scores indicating increased fatigue
The Feeling Scale - Pre-exercise | Immediately before each exercise session
  11 point scale of perceived affect during exercise, positive scores indicating positive affect, negative scores indicating negative affect
The Feeling Scale - Post-exercise | Immediately after each exercise session
  11 point scale of perceived affect during exercise, positive scores indicating positive affect, negative scores indicating negative affect
Rate of perceived exertion | Immediately after every exercise session
  11 point scale of perceived work/intensity during exercise. Higher scores indicate more intense workout.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Marker, PT, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Anschutz Health and Wellness, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marker RJ, Kittelson AJ, Scorsone JJ, Moran IA, Quindry JC, Leach HJ. A Novel Telehealth Exercise Program Designed for Rural Survivors of Cancer With Cancer-Related Fatigue: Single-Arm Feasibility Trial. JMIR Cancer. 2025 Jan 10;11:e59478. doi: 10.2196/59478. PMID 39793972